CLINICAL TRIAL: NCT00101010
Title: A Phase II Study Of Rituximab-CHOP With Pegylated Liposomal Doxorubicin In Patients Older Than 60 Years Of Age With Untreated Aggressive B-Cell Non-Hodgkin's Lymphoma
Brief Title: Rituximab and Combination Chemotherapy in Treating Older Patients With Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000407533; MDA-CCOP-2004-0305; NCI-6485; 2004-0305 (Other: UT MD Anderson Cancer Center); NCI-2009-00064 (Registry Identifier: NCI CTRP); 2U10CA045809 (NIH); NCT00290446 (obsolete NCT alias)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; pegylated granulocyte colony-stimulating factor, human; Rituximab; Cyclophosphamide; liposomal doxorubicin; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab - Combination Chemotherapy (Experimental): Rituximab 375 mg/m^2 intravenous (IV), Cyclophosphamide IV over 1-1½ hours, Pegylated doxorubicin HCl liposome 40 mg/m^2 IV over 1 hour, Vincristine 2 mg IV, day 1, & oral Prednisone 40 mg/m^2 days 1 - 5; Filgrastim (G-CSF) 5 mcg/kg subcutaneously (SC) once daily beginning day 6 continuing until blood counts recover OR Pegfilgrastim 6 mg SC once on day 6 (24 hours after chemotherapy). Treatment repeats every 21 days for up to 8 courses.
  Interventions: Biological: Filgrastim; Biological: Pegfilgrastim; Biological: Rituximab; Drug: Cyclophosphamide; Drug: Pegylated liposomal doxorubicin hydrochloride; Drug: Prednisone; Drug: Vincristine Sulfate

INTERVENTIONS:
Biological: Filgrastim — 5 mcg/kg, SC daily, start 24 hours after chemotherapy
  Other Names: G-CSF; Neupogen
Biological: Pegfilgrastim — 6 mg SC one time (24 hours after chemotherapy)
  Other Names: Neulasta; PEG-G-CSF
Biological: Rituximab — 375 mg/m^2 intravenous piggy back (IVPB) on day 1, administered 1st
  Other Names: Rituxan
Drug: Cyclophosphamide — 750 mg/m^2 IVPB on day 1
  Other Names: Cytoxan; Neosar
Drug: Pegylated liposomal doxorubicin hydrochloride — 40 mg/m^2 IV (maximum dose 90 mg) infusion over 1 hour on day 1
  Other Names: Caelyx; Doxil; liposomal doxorubicin; doxorubicin hydrochloride; liposomal doxorubicin hydrochloride
Drug: Prednisone — 40 mg/m^2 oral days 1 - 5.
Drug: Vincristine Sulfate — 2 mg IV, day 1

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with combination chemotherapy works in treating older patients with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response rate in older patients with previously untreated aggressive diffuse large B-cell stage II-IV lymphoma treated with rituximab, cyclophosphamide, pegylated doxorubicin hydrochloride liposome (HCl), vincristine, and prednisone.
* Determine the cardiotoxicity and myelosuppression of this regimen in these patients.

Secondary

* Determine disease-free survival and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive rituximab intravenous (IV), cyclophosphamide IV over 1-1½ hours, pegylated doxorubicin HCl liposome IV over 1 hour, and vincristine IV on day 1, and oral prednisone on days 1-5. Patients also receive filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 6 and continuing until blood counts recover OR pegfilgrastim SC once on day 6 (24 hours after the completion of chemotherapy). Treatment repeats every 21 days for up to 8 courses in the absence of unacceptable toxicity, disease progression, active hepatitis B virus infection, or hepatitis. Patients with no response OR who achieve less than a partial response after 4 courses are removed from the study.

Patients are followed at 1 month, every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A maximum of 80 patients will be accrued for this study within 27 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diffuse large B-cell lymphoma

  * Stage II, III, or IV disease
  * Previously untreated disease
* Measurable or evaluable disease
* No primary central nervous system (CNS) lymphoma or follicular B-cell lymphoma

PATIENT CHARACTERISTICS:

Age

* 61 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3*
* Platelet count > 100,000/mm^3* NOTE: * Unless due to lymphoma-related hypersplenism or bone marrow infiltration

Hepatic

* Bilirubin < 2 mg/dL
* Hepatitis B surface antigen negative
* Hepatitis B core antibody negative
* Hepatitis C Virus antibody negative

Renal

* Creatinine < 2 mg/dL

Cardiovascular

* left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram or ple gated acquisition (MUGA) scan
* No uncontrolled hypertension or cardiac symptoms
* Cardiologist consultation required for patients with stage A cardiac failure or any of the following known heart diseases:

  * Diastolic dysfunction
  * Prior coronary artery bypass graft
  * Prior percutaneous transluminal coronary angioplasty
  * Prior stent insertion
  * Prior radiotherapy to the chest
* No myocardial infarction within the past 6 months
* No New York Heart Association class II-IV heart failure
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No clinically significant pericardial disease
* No acute ischemic or active conduction system abnormality by electrocardiogram (EKG)

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No psychiatric illness that would preclude study compliance or giving informed consent
* No other major life-threatening illness that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Cardiovascular

Surgery

* See Cardiovascular

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria A. Rodriguez, MD, Study Chair — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Cancer Research for the Ozarks, Springfield, Missouri
  - Hematology Oncology Associates of Central New York, PC - Northeast Center, East Syracuse, New York
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Texas M.D. Anderson CCOP Research Base, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab - Combination Chemotherapy
Started | 80
Completed | 79
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab - Combination Chemotherapy
Number analyzed (Participants) | 80
Age, Customized [Number; unit: participants]
  60 to 69 | 40
  70 to 79 | 27
  80 to 89 | 12
  90 to 99 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Disease Response (Complete, Complete Unconfirmed, and Partial Responses) After 4 Courses
Description: Response was defined as participants with a complete response (CR), unconfirmed complete response (CRu) or partial response (PR), based on International Workshop Criteria (IWG) for Tumor Response Criteria assessed with CT & FDG-PET scans at 4 cycles (12 weeks). CR defined as disappearance of all target and non-target lesions in liver & spleen, & all lymph node masses regressed to normal size. PR defined as ≥50% reduction in sum of product of diameters (SPD) for measured lymph nodes, splenic & liver lesions separately compared to baseline SPD. CRu does not qualify for CR above, due to a residual nodal mass or an indeterminate bone marrow.
Time Frame: Evaluation after 12 weeks (4 cycles of 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab - Combination Chemotherapy
Number analyzed (Participants) | 79
Participants
  Complete Response (CR) | 47
  Uncomfirmed Complete Response (CRu) | 8
  Partial Response (PD) | 14

2. Primary Outcome: Number of Participants Experienced Grade 3 or Higher Cardiac Toxicity After Treatment: Cardiac Toxicity as Measured by Left Ventricular Ejection Fraction (LVEF) on Echocardiogram (ECHO) After 8 Courses
Description: Ejection fraction ( EF) refers to the amount, or percentage, of blood that is pumped (or ejected) out of the ventricles with each contraction. Cardiology evaluation performed before second dose of pegylated liposomal doxorubicin or before entry onto trial, re-evaluation by cardiologist obtained in asymptomatic patients after chemotherapy cycle 4 and again after completion of therapy, and more often if symptomatic. Severe cardiac toxicity considered to be both Grade 3 and 4, and are graded according to NCI common toxicity criteria, CTCAE version 3.0.
Time Frame: Up to 24 weeks (8 cycles of 21 days)
Measure: Number; unit: participants
Arm/Group | Rituximab - Combination Chemotherapy
Number analyzed (Participants) | 80
participants | 10

3. Secondary Outcome: Survival Rate
Description: The percentage of participants still alive after treatment. Survival information obtained 1 month after completion of treatment, then every 3 months for 1 year, every 4 months for one year and every 6 months thereafter.
Time Frame: Up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Disease-free Survival
Description: The percentage of participants with no disease progression for period of time after treatment. Survival assessed every 3 months for 1 year, every 4 months for 2 years, every 6 months for 3 years, and then yearly thereafter up to 5 years.
Time Frame: Up to 5 years or until disease progression
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event collection from first of treatment up to completion of eight cycles of 21 days, approximately 24 weeks.
Arm/Group | Rituximab - Combination Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/80
Other Adverse Events (participants affected / at risk) | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab - Combination Chemotherapy (N=80)
LEPTOMENINGEAL (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No